CLINICAL TRIAL: NCT06283498
Title: Transvaginal Detrusor Nerve Radiofrequency Ablation for Treatment of Overactive Bladder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO612574A
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Treatment (Experimental): 20 female patients with overactive bladder symptoms, aged 21 to 80 years old, inclusive from two sites.
  Interventions: Device: Device Morpheus8V

INTERVENTIONS:
Device: Device Morpheus8V — Assigned to be treated using the modified Morpheus8V

SUMMARY:
The goal of this Safety and efficacy of transvaginal Detrusor Nerve Ablation for treatment of overactive bladder symptoms, including refractory overactive bladder

The main questions it aims to answer are:

•Change from baseline to the end of treatment in a 3-day diary analysis to assess the reduction of urgency incontinence episodes. [Time Frame: 3 months]

Subjects will undergo one treatment session and be reassessed at 4 weeks post-treatment. If less than a 50% improvement is noted, a second and third treatment session will be performed at 4-week intervals. If more than a 50% improvement is noted, patients will be followed longitudinally to assess the durability of the treatment. Investigators will have the ability to initiate a second and or third treatment on an individual basis.

Follow-up will occur at 3- months, 6-months and 12 months after the subject's last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years old, inclusive
* Subject is willing to provide Informed Consent, is geographically stable, understands the requirements for completing the bladder diary and is willing to comply with the required diary, follow-up visits, and testing schedules.
* Urinary incontinence, predominant urgency incontinence for at least one episode on a 3-days diary.
* Reporting at least "moderate bother" on Item 2 on the UDI, "Do you experience a strong feeling of urgency to empty your bladder" (on new patient paperwork)
* >8 micturitions and >3 urgency episodes per 24 hours on a 3-day bladder diary (see Appendix 2)
* 1 UUI episode on a 3-day bladder diary (see Appendix 2)
* Not currently taking anti-muscarinic or beta3 agonist therapy (after at least a 2-week wash-out period)
* Post-void residual (PVR) ≤ 100 ml NOTE: it may include Subjects with a single PVR of >100 ml followed by two consecutive PVR measurements of ≤100 ml in the study. We will record the final acceptable PVR measurement in the data.
* Ability and willingness to self-catheterize in case this is necessary.
* With respect to their reproductive capacity must be post-menopausal or surgically sterile or willing to use a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly from screening until the last follow up

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other metallic or electronic implant anywhere in the body.
* Any permanent implant or an injected chemical substance in the treatment area.
* Superficial areas that have been injected with HA/collagen/fat injections or other augmentation methods with bio-material during last 6 months.
* Current or history of cancer, or current condition of any other type of cancer, or premalignant moles.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy, the intention of pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, autoimmune disorders, or use of immunosuppressive medications.
* Patients with a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction and hormonal virilization.
* Any active condition in the treatment area, such as sores, eczema, and rash.
* History of vaginal disorders, keloids, abnormal wound healing.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days, as per the practitioner's discretion.
* Non-English speakers
* Severely impaired mobility or cognition
* Spinal cord injury or advanced/severe neurologic condition including Multiple Sclerosis, Parkinson's Disease
* Repair of pelvic organ prolapse or incontinence procedure in the previous 6 months
* Ongoing complications of prior anti-incontinence surgery
* Received intravesical botulinum injection within the previous 12 months
* History of an implanted nerve stimulator for incontinence
* History of prior sling or vaginal mesh placement,
* Previous diagnosis of interstitial cystitis, bladder cancer, or chronic pelvic pain
* Current participation in any other conflicting interventional or OAB treatment study
* Planning to become pregnant during the study period.
* Pelvic radiation, history of pelvic radiation
* Subject with 24-hour total urine volume voided greater than 3,000 ml as measured at screening period.
* Active urinary tract or vaginal infection
* Anatomical conditions that would prevent the introduction and use of the device, in such as significant pelvic organ prolapse,
* Current hydronephrosis or hydroureter
* Bladder outflow obstruction
* Active pelvic organ malignancy
* Urethral obstruction
* Urinary retention or prolonged catheter use
* Less than 12 months post-partum or currently pregnant or plan to become pregnant in the following 12 months.
* Untreated symptomatic urinary tract infection
* Unevaluated hematuria
* Medical instability
* Allergy to anesthetics as Benzocaine/Lidocaine/Tetracaine Cream (BLT Cream) used in the study
* Not available for follow-up in 6 months
* Participation in other research trials that could influence results of this study

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20 female patients with overactive bladder symptoms, aged 21 to 80 years old, inclusive from two sites .
Enrollment: 32 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Change in urgency incontinence episodes after 3 month | 3 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the reduction of urgency incontinence episodes.

SECONDARY OUTCOMES:
Change in urgency incontinence episodes after 1 month | 1 month
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the reduction of urgency incontinence episodes
Change in urgency incontinence episodes | 6 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the reduction of urgency incontinence episodes.
Change in urgency incontinence episodes | 12 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the reduction of urgency incontinence episodes.
Analysis to assess the urinary frequency | 1 month
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the urinary frequency.
Analysis to assess urinary frequency | 3 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess urinary frequency.
Analysis to assess the urinary frequency. | 6 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the urinary frequency. [Time Frame: 6 months]
Analysis to assess the urinary frequency. | 12 months
  Change from baseline to the end of treatment in a 3-day diary analysis to assess the urinary frequency.
Assessment of the impact of the treatment on Overactive Bladder symptoms | 1 month
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Assessment of the impact of the treatment on Overactive Bladder symptoms | 3 months
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Assessment of the impact of the treatment on Overactive Bladder symptoms | 6 months
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Assessment of the impact of the treatment on Overactive Bladder symptoms | 12 months
  Measured by the Incontinence Impact Questionnaire Total Score. Normative values for a general population, 10% of whom scored above 4.8 on IIQ-7. Values obtained from patients with severe incontinence indicate that a score > 70 on the IIQ signifies a poor QOL. Lower scores on IIQ-7 may identify more females who are bothered by urinary incontinence. 7 items are divided into four domains (physical activity, travel, social relationships, emotional health). Item-level scores are rated on a four-point Likert scale (where 0=not at all and 3=greatly), determined by the self-reported impact of symptoms related to urinary incontinence.
  The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Patient-reported Pain assessment | treatment procedure
  The subject will be asked to rate the severity from 0 to 10, with 0 equaling no symptoms and 10 equaling the worst possible symptoms. A number is obtained by measuring up to the point the subject has indicated.
Patient-reported outcome measure | 1 month
  Patient perception of bladder condition and device acceptance measured by Patient Satisfaction Questionnaire. 6 points Likert scale, grading from 0 to 5. A lower score indicates a better outcome.
Patient-reported outcome measure | 3 months
  Patient perception of bladder condition and device acceptance measured by Patient Satisfaction Questionnaire. 6 points Likert scale, grading from 0 to 5. A lower score indicates a better outcome.
Patient-reported outcome measure | 6 months
  Patient perception of bladder condition and device acceptance measured by Patient Satisfaction Questionnaire. 6 points Likert scale, grading from 0 to 5. A lower score indicates a better outcome.
Patient-reported outcome measure | 12 months
  Patient perception of bladder condition and device acceptance measured by Patient Satisfaction Questionnaire. 6 points Likert scale, grading from 0 to 5. A lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mickey Karram, MD, Principal Investigator — Not Affiliated
Locations (3):
- United States (2):
  - Mickey Karram MD, Corona del Mar, California
  - Institute for Female Pelvic Medicine, Knoxville, Tennessee
- The Hospital Infantil Universitario de San José (University Children's Hospital of San José), Bogotá, Colombia